CLINICAL TRIAL: NCT04040894
Title: Phase 3b, Multicenter, Open-label, Single-Arm Expanded Access Protocol of TEPROTUMUMAB (HZN-001)
Brief Title: Expanded Access Protocol of Teprotumumab (HZN-001) for Patients With Active Thyroid Eye Disease
Acronym: EAP
Status: Approved for marketing | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: HZNP-TEP-401
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Thyroid Eye Disease; Graves' Orbitopathy
Keywords: Proptosis; Human monoclonal antibody; insulin-like growth factor-1 receptor; Thyroid-Associated Ophthalmopathy; Hyperthyroidism; Autoimmune Thyroid Disease
MeSH Terms: conditions — Graves Ophthalmopathy; Exophthalmos; Hyperthyroidism | interventions — teprotumumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Teprotumumab — Treatment with 8 infusions of Teprotumumab q3W for a total of 21 weeks. Teprotumumab 10 mg/kg will be administered on Day 1 and Teprotumumab 20 mg/kg will be administered q3W for the remaining 7 infusions.
  Other Names: HZN-001

SUMMARY:
This is an expanded access protocol intended to provide access to teprotumumab for the treatment of up to 60 patients in the United States with active moderate to severe thyroid eye disease where there is no comparable or satisfactory alternative therapy for treatment.

DETAILED DESCRIPTION:
Requests for access to the Sponsor must be made by a licensed physician for a specific patient, based on a determination with the patient that the benefits of treatment with the investigational drug outweigh the risks. Licensed physician's with eligible patients must apply and meet requirements for participation in the expanded access program.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female patient at least 18 years old.
3. Clinical diagnosis active TED with a CAS ≥ 4 (on the 7-item scale).
4. Moderate-to-severe active TED (not sight-threatening but has an appreciable impact on daily life), usually associated with one or more of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, exophthalmos ≥ 3 mm above normal for race and gender, and/or inconstant or constant diplopia.
5. Onset of Active TED symptoms (as determined by patient records) within approximately 12 months prior to eligibility review.
6. Patients must be euthyroid with the baseline disease under control or have mild hypo- or hyperthyroidism (defined as free thyroxine [FT4] and free triiodothyronine [FT3] levels < 50% above or below the normal limits) at Eligibility review. Every effort should be made to correct the mild hypo- or hyperthyroidism promptly and to maintain the euthyroid state for the full duration of participation.
7. Does not require immediate surgical ophthalmological intervention.
8. Diabetic patients must have well-controlled stable disease (defined as HbA1c < 9.0%).
9. Women of childbearing potential (including those with an onset of menopause <2 years, non-therapy-induced amenorrhea for <12 months, or not surgically sterile [absence of ovaries and/or uterus]) must have a negative serum pregnancy test within 3 weeks prior to the first infusion and negative urine pregnancy tests at all protocol-specified timepoints (i.e., prior to each infusion); patients who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the expanded access program, one of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started at least one full cycle prior to the first infusion and continue for 180 days after the last dose of investigational drug. Highly effective contraceptive methods (with a failure rate less than 1% per year), when used consistently and correctly, includes implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner.
10. Male patients must be surgically sterile or, if sexually active with a female partner of childbearing potential, must agree to use a barrier contraceptive method from the first infusion through 180 days after the last dose of investigational drug.
11. Patient is willing and able to comply with the prescribed treatment protocol and evaluations for the duration of their participation.

Exclusion Criteria:

1. Any treatment with rituximab (Rituxan® or MabThera®) within 12 months prior to the first infusion of teprotumumab or tocilizumab (Actemra® or Roactemra®) within 6 months prior to the first infusion of teprotumumab. Use of any other non-steroid immunosuppressive agent within 3 months prior to the first infusion of teprotumumab.
2. Use of an investigational agent for any condition within 60 days prior to the first infusion or anticipated use during the course of the protocol.
3. Pregnant or lactating women.
4. Biopsy-proven or clinically suspected IBD (e.g., diarrhea with or without blood or rectal bleeding associated with abdominal pain or cramping/colic, urgency, tenesmus, or incontinence for more than 4 weeks without a confirmed alternative diagnosis OR endoscopic or radiologic evidence of enteritis/colitis without a confirmed alternative diagnosis).
5. Known hypersensitivity to any of the components of teprotumumab or prior hypersensitivity reactions to mAbs.
6. Any other condition that, in the opinion of the Sponsor, would preclude inclusion in the expanded access program.
7. Previous enrollment in this study or participation in a prior teprotumumab clinical study.
8. Human immunodeficiency virus, hepatitis C or hepatitis B infections.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (8):
  - MACRO Trials, Beverly Hills, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - NorthShore University HealthSystem, Skokie, Illinois
  - Institute of Ophthalmology and Visual Science, Rutgers University New Jersey Medical School, Newark, New Jersey
  - Eye and Facial Plastic Surgery Consultants, Plymouth Meeting, Pennsylvania
  - Prisma Health Upstate/Endocrinology Specialists and Thyroid Center, Greenville, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - TN Oculoplastics, Nashville, Tennessee

REFERENCES:
- See also: Related Info — http://tepezza.com